CLINICAL TRIAL: NCT06882941
Title: Modulation of the Gut Microbiota and Metabolism in Elderly by Algae Products.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 201804003RINB
Record Dates: First submitted 2025-01-07; First posted 2025-03-19 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2018-05

CONDITIONS: Frailty
Keywords: frailty; Black soybean; Adlay; fermentation; gut microbiota
MeSH Terms: conditions — Frailty

STUDY DESIGN:
Intervention Model Description: Parcitipants will be stratified randomization into placebo and experimental groups based on their robustness status.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Non-Fermented Black Soybean and Adlay Supplement (Placebo Comparator): The placebo product was prepared using uninoculated autoclaved black soybean and dehulled adlay. The samples were provided as frozen food and required microwaving for 30 seconds before serving. Participants assigned to the placebo group will take the non-fermented black soybean and adlay supplement daily for 12 weeks.
  Interventions: Dietary Supplement: non-fermented black soybean and adlay supplement
- Fermented Black Soybean and Adlay Supplement (Experimental): The preparation of the fermented black soybean and adlay supplement involves autoclaved black soybean and dehulled adlay, which are inoculated with Bacillus subtilis natto (1.3 × 10⁶ CFU/g) and incubated for 43 hours at 28°C. Participants assigned to the experimental group will take the Fermented Black Soybean and Adlay Supplement daily for 12 weeks.
  Interventions: Dietary Supplement: Fermented Black Soybean and Adlay Supplement

INTERVENTIONS:
Dietary Supplement: Fermented Black Soybean and Adlay Supplement — The preparation of the fermented black soybean and adlay supplement involves autoclaved black soybean and dehulled adlay, which are inoculated with Bacillus subtilis natto (1.3 × 10⁶ CFU/g) and incubated for 43 hours at 28°C. Participants assigned to the experimental group will take the Fermented Black Soybean and Adlay Supplement daily for 12 weeks.
  Arms: Fermented Black Soybean and Adlay Supplement
Dietary Supplement: non-fermented black soybean and adlay supplement — The placebo product was prepared using uninoculated autoclaved black soybean and dehulled adlay. The samples were provided as frozen food and required microwaving for 30 seconds before serving. Participants assigned to the placebo group will take the non-fermented black soybean and adlay supplement daily for 12 weeks.
  Arms: Non-Fermented Black Soybean and Adlay Supplement

SUMMARY:
The goal of this clinical trial is to determine whether a fermented black soybean and adlay supplement can improve frailty. The main questions it seeks to answer are:

* Does the fermented black soybean and adlay supplement improve physical performance?
* What is the effect of the fermented black soybean and adlay supplement on gut microbiota? Researchers will compare the fermented black soybean and adlay supplement to a placebo (a non-fermented black soybean and adlay supplement) to assess its impact on physical performance.

Participants will:

* Take either the fermented black soybean and adlay supplement or a placebo daily for 12 weeks.
* Visit the clinic for checkups and tests before and after consuming the product.

DETAILED DESCRIPTION:
This study aims to evaluate the effects of fermented black soybean and adlay supplements on frailty and gut microbiota in older adults. Older participants are recruited from National Taiwan University Hospital. Parcitipants will be stratified randomization into placebo and experimental groups based on their robustness status. Older participants will take either the fermented black soybean and adlay supplement or a placebo daily for 12 weeks. Baseline characteristics of the participants, including demographic data, chronic disease history, and anthropometric data, will be collected. Cognitive function will be evaluated using the Mini-Mental Status Examination. A 15-item version of the Geriatric Depression Scale will be used to identify depressive symptoms. Nutritional status will be assessed with the Mini Nutritional Assessment. Blood and fecal samples, as well as data on physical performance and frailty status, will be collected before and after consuming the product.

ELIGIBILITY:
Inclusion Criteria:

* Age 65 years or older
* Independent in activities of daily living

Exclusion Criteria:

* Being bedridden or residing in a nursing home
* Having a life expectancy of less than 6 months
* Having severe hearing or communication disorders
* Having hyperuricemia, gouty arthritis, or swallowing dysfunction

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 141 (Actual)
Dates: Start 2018-12-12 (Actual); Primary Completion 2020-12-17 (Actual); Study Completion 2021-04-16 (Actual)

PRIMARY OUTCOMES:
frailty status | From enrollment to the end of treatment at 12 weeks
  Frailty status will be assessed using modified Fried's criteria before and after consuming the product.

SECONDARY OUTCOMES:
gut microbiota | From enrollment to the end of treatment at 12 weeks
  Gut microbiota will be analyzed via fecal sample collection before and after consuming the product.
Physical performance: 5-meter walk speed | From enrollment to the end of treatment at 12 weeks
  5-meter walk speed will be evaluated before and after consuming the product. The participant will be asked to walk at their normal comfortable pace until they reach the end of the 5-meter mark.
physical performance: Timed Up and Go test | From enrollment to the end of treatment at 12 weeks
  Timed Up and Go test will be evaluated before and after consuming the product. The Timed Up and Go test measures functional mobility by timing a participant as they rise from a chair, walk 3 meters, turn around, walk back, and sit down.
physical performance: 30-second chair stand test | From enrollment to the end of treatment at 12 weeks
  Thirty-second chair stand test will be evaluated before and after consuming the product.
  The 30-Second Chair Stand Test measures lower body strength and endurance by counting the number of times a participant can fully stand up from a chair and sit back down within 30 seconds.
physical performance: grip strength | From enrollment to the end of treatment at 12 weeks
  Grip strength will be measured before and after consuming the product. Grip strength measurement assesses upper body muscle strength by using a dynamometer to measure the maximum force exerted when a participant squeezes the device with their dominant hand.
Number of participants with biochemistry blood tests. | From enrollment to the end of treatment at 12 weeks
  Biochemical data from blood samples of the 141 participants will be analyzed before and after consuming the product.

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No